CLINICAL TRIAL: NCT03112746
Title: Efficacy of the Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach With Brazilian Children With Developmental Coordination Disorder
Brief Title: Efficacy of the CO-OP Approach With Brazilian Children With Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Clarice Ribeiro Soares Araujo, Master in Rehabilitation Sciences, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COEP/UFMG ETIC Nº 103/2009
Record Dates: First submitted 2017-04-02; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Developmental Coordination Disorder
Keywords: child; goal; intervention; motor skills disorder; occupational therapy
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Orientation to daily Occupational Performance (Experimental): One group was submitted to the CO-OP approach to learn cognitive strategies to perform the chosen tasks.
  Interventions: Behavioral: Cognitive Orientation to Daily Occupational Performance

INTERVENTIONS:
Behavioral: Cognitive Orientation to Daily Occupational Performance — In CO-OP Approach, therapists use mediational techniques to teach cognitive strategies - GOAL, PLAN, DO, CHECK - to improve occupational performance in goals chosen by the children in collaboration with them and their parents.
  Other Names: CO-OP Approach

SUMMARY:
Children with Developmental Coordination Disorder (DCD) have difficulties performing daily activities which reflects negatively on participation, impacting their lives. To date, there are a number of interventions to improve performance of these children on activities they want or need to. In Brazil, there is little research on the efficacy of such approaches. Our main objective was to start a set of studies to examine the effects of the Cognitive Orientation to Daily Occupational Performance Approach (CO-OP Approach) protocol on occupational performance and satisfaction of Brazilian children who have DCD; to examine whether children were able to transfer strategies and skills learned during CO-OP to untrained goals.

DETAILED DESCRIPTION:
Background. Children with Developmental Coordination Disorder (DCD) have difficulties performing daily activities which reflects negatively on participation, impacting their lives. Objectives. To examine the effects of the Cognitive Orientation to Daily Occupational Performance Approach (CO-OP Approach) protocol on occupational performance and satisfaction of Brazilian children who have DCD; to examine whether children were able to transfer strategies and skills learned during CO-OP to untrained goals. Methods. A pre-post group comparison design with eight boys aged 6-10 years old. Children participated in 12 CO-OP sessions with their parents twice a week, with an extra session added to the protocol for parents´ orientation. The Canadian Occupational Performance Measure and the Performance Quality Rating Scale were used as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* poor motor performance measured by a motor performance test (cut off score below the 15th percentile).
* poor performance on academic and daily living activities measured by the Developmental Coordination Disorder Questionnaire answered by the parents.
* attending regular education with no evidence of marked school delay (over a year).
* cognitive development within the expected age range according to the Wechsler Intelligence Scale for Children-Third Edition (WISC-III).

Exclusion Criteria:

* signs of neurological or neuromuscular disorder.
* presence of intellectual disability.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2009-03-26 (Actual); Primary Completion 2010-02-10 (Actual); Study Completion 2010-03-26 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | up to 12 weeks
  Change on performance and satisfaction on goals chosen by each child
Performance Quality Rating Scale | up to 12 weeks
  Change on occupational performance on goals chosen by each child as measured by external evaluators

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller LT, Polatajko HJ, Missiuna C, Mandich AD, Macnab JJ. A pilot trial of a cognitive treatment for children with developmental coordination disorder. Hum Mov Sci. 2001 Mar;20(1-2):183-210. doi: 10.1016/s0167-9457(01)00034-3. PMID 11471396
- [Background] Mandich AD, Polatajko HJ, Macnab JJ, Miller LT. Treatment of children with Developmental Coordination Disorder: what is the evidence? Phys Occup Ther Pediatr. 2001;20(2-3):51-68. PMID 11345512
- [Background] Mandich AD, Polatajko HJ, Rodger S. Rites of passage: understanding participation of children with developmental coordination disorder. Hum Mov Sci. 2003 Nov;22(4-5):583-95. doi: 10.1016/j.humov.2003.09.011. PMID 14624835
- [Background] Green D, Chambers ME, Sugden DA. Does subtype of developmental coordination disorder count: is there a differential effect on outcome following intervention? Hum Mov Sci. 2008 Apr;27(2):363-82. doi: 10.1016/j.humov.2008.02.009. Epub 2008 Apr 8. PMID 18400322
- [Background] Carswell A, McColl MA, Baptiste S, Law M, Polatajko H, Pollock N. The Canadian Occupational Performance Measure: a research and clinical literature review. Can J Occup Ther. 2004 Oct;71(4):210-22. doi: 10.1177/000841740407100406. PMID 15586853
- [Derived] Araujo CRS, Cardoso AA, Magalhaes LC. Efficacy of the cognitive orientation to daily occupational performance with Brazilian children with developmental coordination disorder. Scand J Occup Ther. 2019 Jan;26(1):46-54. doi: 10.1080/11038128.2017.1417476. Epub 2017 Dec 20. PMID 29260603